CLINICAL TRIAL: NCT03504787
Title: Upper Extremity Selective Voluntary Motor Control in Children With Unilateral Cerebral Palsy and Its Association With Upper Extremity Function
Brief Title: Upper Extremity Selective Voluntary Motor Control in Children With Unilateral Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayse Simsek, Research assistant, Gazi University
Other Study IDs: 77082166-302.08.01
Record Dates: First submitted 2018-04-10; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; upper extremity; selective motor control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to determine upper extremity selective motor control (SMC) in Children with Unilateral Cerebral Palsy (CP). It was also aimed to determine the relationship between upper extremity SMC and upper extremity functions in unilateral CP.

DETAILED DESCRIPTION:
Twenty-four unilateral CP participated in the study between the ages of 6 and 18 years. Children's manual skills classified with MACS. To assess the quality of the upper extremity, the Quality of Upper Extremity Skill Test (QUEST) which assessed four areas including dissociated movement, grasp, weight bearing and protective extension, was used. Upper extremity functions were assessed using the Jebsen Taylor Hand Function Test (JTT). The Selective Control of Upper Extremity Scale (SCUES) was used to evaluate the selective movements of the upper extremity. The SCUES evaluates the movement of the trunk during the upper limb movements and mirror movements via video recording.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of unilateral spastic CP,
* age between 5 and 18 years,
* ability to follow simple instructions.

Exclusion Criteria:

* significant ataxia or dystonia
* orthopedic intervention or botulinum toxin injection to the upper extremities in the last 6 months
* orthopedic problems or medical conditions that prevented children from participating in the assessment

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with unilateral cerebral palsy.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-03-25 (Actual)

PRIMARY OUTCOMES:
Selective Control of the Upper Extremity Scale (SCUES) | 10 minutes
  The SCUES evaluate for movement at each joint level: the presence of mirror movements, movement of additional joints the target or index joint, presence of trunk movement, dynamic motion less than passive ROM. Upper extremity joint levels and motions examined include the shoulder (abduction/adduction), elbow (flexion/extension), forearm (supination/pronation), wrist (flexion/extension), and fingers/thumb (grasp/release). A video camera is placed in front of a participant sitting on a table. The examiner demonstrate the desired motion to the participant, then passively moves the participant's joint in the desired planes. The participant is then asked to perform the same motion. This activity is graded by the examiner from the videotape. Evaluation lasts less than 15 minutes. Motion at each of the five joint levels is graded on a four-point scale: no SMC, moderately diminished SMC, mildly diminished SMC, and normal SMC

SECONDARY OUTCOMES:
Jebsen Taylor Hand Function Test (JTT) | 10 minutes
  It is a standard test used to evaluate the general hand function of the person. Seven subsets of the test simulate hand function, which includes writing, simulated page turning, stacking checkers, simulated feeding and picking up small common objects, large light objects, large heavy objects
Quality of Upper Extremity Skill Test (QUEST) | 20 minutes
  The QUEST evaluates the quality of the upper extremity to four areas; Dissociated Movement, Grasp, Weight Bearing and Protective Extension. A score of "yes" or "no" is given according to the completion of each movement or task. The four field scores are summed to achieve the total score. During evaluation, the child is not allowed to use any device in the upper extremity

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Elbasan, Study Chair — Gazi University
Locations (1):
- Gazı University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No